CLINICAL TRIAL: NCT01004783
Title: Validation of Prognostic Markers for Very Low Risk Wilms Tumors
Brief Title: Biomarkers in Tumor Tissue Samples From Young Patients With Very Low Risk Wilms Tumors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN10B1; COG-AREN10B1 (Other: Children's Oncology Group); CDR0000657973 (Other: Clinical Trials.gov); NCI-2011-02199 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Cancer
Keywords: stage I Wilms tumor; stage II Wilms tumor; epithelial predominant Wilms tumor
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — DNA Methylation; Gene Expression Profiling; Microarray Analysis; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Genetic: loss of heterozygosity analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This clinical trial studies biomarkers in tumor tissue samples from young patients with very low risk Wilms tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To validate the utility of CUGBP2, HMGA2, and MEIS2 mRNA expression and 11p15 methylation to define a population of pediatric patients with very low risk Wilms tumor (VLRWT) that have virtually no risk of relapse.
* To validate the utility of WT-1 mutation and 11p15 loss of heterozygosity analysis to determine a population of VLRWT that have a higher risk of relapse when not treated with chemotherapy.
* To validate the utility of NFYA, STRA6, TOB2, PDCD4, and SP3 mRNA expression to predict relapse in VLRWT.
* To investigate the feasibility of broadening the definition of VLRWT through analysis of stage I and II epithelial differentiated tumors registered on clinical trial COG-Q9401 (NWTS-5) for CUGBP2, HMGA2, MEIS2, and 11p15 methylation.

OUTLINE: Previously banked tumor tissue samples are analyzed for mRNA expression of CUGBP2, HMGA2, and MEIS2 via reverse-transcriptase (RT)-PCR and are classified as loss of heterozygosity (LOH), loss of imprinting, or neither via 11p15 analysis. Samples are also analyzed for WT-1 mutation via quantitative PCR and 11p LOH using 11p15 methylation analysis and expression of NFYA, STRA6, TOB2, PDCD4, and SP3 via quantitative RT-PCR

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patient with very low risk Wilms tumor registered on clinical trial COG-AREN03B2
  * Patient with stage I or II epithelial tubular differentiated Wilms tumor registered on clinical trial COG-Q9401 (NWTS-5)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not Specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with very low risk Wilms tumor registered on clinical trial COG-AREN03B2 or patients with stage I or II epithelial tubular differentiated Wilms tumor registered on clinical trial COG-Q9401 (NWTS-5)
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Utility of CUGBP2, HMGA2, and MEIS2 mRNA expression and 11p15 methylation to define a population of pediatric patients with very low risk Wilms tumor (VLRWT) that have virtually no risk of relapse
Utility of WT-1 mutation and 11p15 loss of heterozygosity analysis to determine a population of VLRWT that have a higher risk of relapse when not treated with chemotherapy
Utility of NFYA, STRA6, TOB2, PDCD4, and SP3 mRNA expression to predict relapse in VLRWT
Feasibility of broadening the definition of VLRWT through analysis of stage I and II epithelial differentiated tumors registered on clinical trial COG-Q9401 (NWTS-5) for CUGBP2, HMGA2, MEIS2, and 11p15 methylation

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. Perlman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago